CLINICAL TRIAL: NCT05593224
Title: The Efficacy and Safety of the Intracranial Stent (Tonbridge) in Endovascular Treatment of Intracranial Atherosclerotic Stenosis: A Prospective, Multicenter, Single-Arm Trial
Brief Title: The Efficacy and Safety of Intracranial Stent (Tonbridge) in Endovascular Treatment of Intracranial Atherosclerotic Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ 202201
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Intracranial Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intracranial Stent (Tonbridge) (Experimental): Placement of Intracranial Stent (Zhuhai Tonbridge Medical Tech. Co., Ltd. ).
  Interventions: Device: Intracranial Stent (Tonbridge)

INTERVENTIONS:
Device: Intracranial Stent (Tonbridge) — The intracranial stent consists of a self-expanding, laser-carved nickel-titanium stent and its delivery system.

SUMMARY:
The purpose of this study is to verify the efficacy and safety of the Intracranial Stent (Tonbridge) in endovascular treatment of intracranial atherosclerotic stenosis.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm clinical trial carried out in 14 centers throughout China. 156 subjects with intracranial atherosclerotic stenosis will be treated with the Intracranial Stent (Tonbridge) for the expansion of vascular stenosis site. The primary objective of this study is to evaluate the effectiveness and safety of the intracranial stent for endovascular treatment of intracranial atherosclerotic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Subjects with symptomatic intracranial atherosclerotic stenosis who do not respond to antiplatelet therapy or have poor compensation of collateral circulation and hypoperfusion in the offending vessel blood supply
* The last onset time of TIA is not limited or the last onset of ischemic stroke is more than 2 weeks
* The lesion is confirmed to be located in intracranial large arteries, including intracranial segment of the internal carotid artery, middle cerebral artery, intracranial segment of vertebral artery and the basilar artery
* Target vessel diameter≥2.0mm and ≤4.5mm, lesion length ≤33mm
* Stenosis degree of intracranial arteries≥70% and ≤99% measured by intracranial angiography (WASID method)
* Intracranial artery stenosis which requiring interventional treatment is a single lesion
* Subjects have at least 1 atherosclerotic plaque risk factor including hypertension, diabetes mellitus, hyperlipidemia, hyperhomocysteinemia, coronary heart disease, obesity, and smoking history
* mRS≤2 before enrollment
* Voluntarily participate in this study and sign the informed consent form, can complete examinations and follow-ups in accordance with the requirements of the protocol during the clinical trial

Exclusion Criteria:

* Intracranial arterial stenosis caused by non-atherosclerotic lesions: such as arterial dissection, moyamoya disease, vasculitis, active arteritis, etc.
* Preoperative MRI shows only perforator infarction in the target lesion
* Preoperative CT or MRI indicates the presence of post-infarct hemorrhagic transformation in the target vascular, or a history of subarachnoid, subdural, and epidural hemorrhage within 30 days before procedure, or the presence of untreated chronic subdural hematoma (≥5mm)
* Severe calcification of target vessels; or target vessel tortuosity or other reasons will make experimental device difficult to reach the target lesion position
* There is more than 70% stenosis in the distal intracranial large vessels or proximal intracranial and extracranial large vessels of the target vessels, and the presence of unidentified responsible lesions
* Subjects have a major surgery within 30 days before procedure or intend to be hospitalized for other procedure within 6 months after procedure
* Intracranial tumors or intracranial arteriovenous malformations, or distal and proximal target vessels combined with aneurysms
* The target lesion has a history of stent implantation
* It is suspected that there is severe allergy or contraindication to aspirin, clopidogrel, heparin, contrast media, nitinol and other drugs and devices related to endovascular therapy
* There is an underlying source of cardiac thrombus, such as atrial fibrillation, left ventricular thrombus, myocardial infarction within 30 days
* Subjects with an INR > 1.5 or the presence of nonmodifiable bleeding factors
* Medically uncontrolled severe hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg)
* Severe comorbid conditions or unstable conditions, such as severe heart failure, pulmonary failure, or renal failure (serum creatinine >3.0 mg/dL (264μmol/L)), severe liver insufficiency (ALT or AST >3 times normal), and malignancy
* Life expectancy is less than two years
* Women who are pregnant or breastfeeding
* Subjects unable to complete follow-up due to cognitive impairment, mood disorder, or mental illness
* Subjects who are enrolled in other clinical trials of drugs/devices and have not yet met the primary endpoint
* Other circumstances which investigators do not consider are appropriate for intracranial stent treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of in-stent restenosis at 6 months | 6 months post-procedure
  The in-stent restenosis is defined as more than 50% stenosis within stent or distal/proximal ends (within 5 mm), and more than 20% absolute lumen loss. The degree of intracranial artery stenosis are measured qualitatively in DSA examination. WASID study will be used to measure the degree of intracranial artery stenosis.

SECONDARY OUTCOMES:
Device success rate and procedural success rate | Intraoperation
  Device success refers to the successful delivery of the stent to the lesion site through the delivery system during procedure, and it is released smoothly and fits well with the vessel wall without bending and displacement; procedural success is defined as stenosis degree less than 30% immediately after procedure.
Incidence of symptomatic in-stent restenosis at 6 months, 1 year, and 2 years | 6 months, 1 year, and 2 years post-procedure
  Symptomatic in-stent restenosis is defined as ischemic stroke or TIA or other ischemic neurological symptoms which are caused by in-stent restenosis.
Ratio of mRS 0-2 at 30 days, 6 months, 1 year, and 2 years | 30 days, 6 months, 1 year, and 2 years post-procedure
  Subjects will be evaluated at the follow-up visits according to the mRS. The mRS 0-2 indicates a good prognosis.
Incidence of stent restenosis at 1 and 2 years | 1 and 2 years post-procedure
  Restenosis is defined as more than 50% stenosis within stent or distal/proximal ends (within 5 mm), and more than 20% absolute lumen loss.
Incidence of any stroke and death within 30 days | Within 30 days post-procedure
  Stroke includes both ischemic and hemorrhagic strokes. Deaths from any cause are included in this data.
Mortality at 31 days to 6 months, 6 to 12 months, and 12 to 24 months | 31 days to 6 months, 6 to 12 months, and 12 to 24 months post-procedure
Incidence of ischemic stroke in the target vessel at 31 days to 6 months, 6 to 12 months, and 12 to 24 months | 31 days to 6 months, 6 to 12 months, and 12 to 24 months post-procedure
Incidence of ischemic stroke in non-target vessel at 31 days to 6 months, 6 to 12 months, and 12 to 24 months | 31 days to 6 months, 6 to 12 months, and 12 to 24 months post-procedure
The incidence of any hemorrhagic stroke at 31 days to 6 months, 6 to 12 months, and 12 to 24 months | 31 days to 6 months, 6 to 12 months, and 12 to 24 months post-procedure
Incidence of device deficiency | After use of device to end of study
  Device deficiency is the unreasonable risk that may endanger human health or life safety in the normal use of medical devices during clinical trials, such as labeling errors, quality problems, malfunctions, etc. Possible device deficiency: labeling errors, product quality problems, design defects, broken sterilization packaging, etc.
Incidence of adverse events (AE) at 30 days, 6 months, 1 year, and 2 years | Through 2 years post-procedure
Incidence of serious adverse events (SAE) at 30 days, 6 months, 1 year, and 2 years | Through 2 years post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital; Shouchun Wang, Principal Investigator — The First Hospital of Jilin University
Locations (14):
- China (14):
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan Science ＆ Technology University, Luoyang, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Baotou City Central Hospital, Baotou, Neimenggu
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Changhai Hospital of Shanghai, Shanghai
  - Tongji Hospitai of Tongji University, Shanghai